CLINICAL TRIAL: NCT03833635
Title: Effects of OMT on Premature Physiological Parameters: a RCT
Brief Title: Effects of OMT on Premature Physiological Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Come Collaboration (Other)
Collaborators: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COME-01-18
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Premature Infant; Physiological Stress
MeSH Terms: conditions — Premature Birth | interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT (Experimental)
  Interventions: Other: osteopathic manipulative treatment
- Control (Placebo Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: osteopathic manipulative treatment — OMT will be used to treat premature infants after having performed a manual osteopathic assessment. Techniques used are indirect
  Arms: OMT
Other: Sham — the sham intervention consists in a stable skin-to-skin contact with the participant
  Arms: Control

SUMMARY:
Osteopathic manipulative treatment has been showed to reduce LOS in premature infants. Despite the clinical effectiveness, lack of data and information on the physiological underpinning effects during the treatment has been revealed. The aim of the study is to explore the immediate physiological effects of osteopathic treatment on premature infants

ELIGIBILITY:
Inclusion Criteria:

* preterm infants

Exclusion Criteria:

* congenital/genetic disease
* cardiovascular/neurological disease

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
heart rate | immediate
  measure of heart rate

SECONDARY OUTCOMES:
oxygen saturation | immediate
  measure of oxygen

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Chieti-Pescara, Chieti
  - Buzzi hospital, Milan

REFERENCES:
- [Derived] Manzotti A, Cerritelli F, Lombardi E, La Rocca S, Chiera M, Galli M, Lista G. Effects of osteopathic treatment versus static touch on heart rate and oxygen saturation in premature babies: A randomized controlled trial. Complement Ther Clin Pract. 2020 May;39:101116. doi: 10.1016/j.ctcp.2020.101116. Epub 2020 Feb 8. PMID 32379655